CLINICAL TRIAL: NCT02304146
Title: Long-term Ultrasound Guided Foam Sclerotherapy Versus Classical Surgical Stripping Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 144144
Record Dates: First submitted 2014-11-11; First posted 2014-12-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Varicose Veins
Keywords: Foam; UGFS; Stripping; Incompetence
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High ligation and stripping (surgery): 6-10 years post classical stripping of the great saphenous vein.
- Foam sclerotherapy: 6-10 years post post ultrasound guided foam sclerotherapy of the great saphenous vein.

SUMMARY:
The aim of this study is to investigate the long-term follow-up of the previously conducted FOAM study.

DETAILED DESCRIPTION:
It describes the long-term quality of life (QoL) after ultrasound guided foam sclerotherapy (UGFS) and surgical stripping, outcomes with regard to clinical, and ultrasound recurrence, progression of venous disease, predictive value of the presence of central / deep venous obstruction for recurrence of varicose veins and the long term cost analysis.

Recurrence of varicose veins was defined as the presence of one or more venous symptoms such as pain, cramps, restless legs and a tired/heavy feeling in the treated leg, in combination with the presence of reflux longer than 0·5 s.

The initial definition of recurrent reflux, which is defined as reflux for more than 2 cm in length in the treated vein segment (proximal great saphenous vein (GSV) ) as measured by colour flow duplex ultrasound (DUS). DUS findings of the treated proximal GSV were categorized as: 1, absence of reflux; 2, reflux; 3, occlusion; 4, partial occlusion with reflux; 5, absence of vein, is being used. Patients in categories 2 and 4 are considered to have reflux.

ELIGIBILITY:
Inclusion Criteria:

* all patients included in previous FOAM study

Exclusion Criteria:

* no received informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were randomized and received the allocated treatment UGFS or surgical stripping.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
long-term QoL follow-up of patients after UGFS and surgical stripping | 6-10 years follow-up

SECONDARY OUTCOMES:
Clinical recurrence | 6-10 years follow-up
Technical recurrence | 6-10 years follow-up
  Vein closure rates
Number of retreatments | 6-10 years follow-up
Venous Clinical Severity Score change | 6-10 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: C.H.A. Wittens, M.D. PhD, Principal Investigator — Maastricht UMC
Locations (3):
- Netherlands (3):
  - Department of Dermatology, Atrium Medical Centre., Heerlen, Limburg
  - Maastricht UMC+, Maastricht, Limburg
  - Departments of Dermatology and Surgery, Laurentius Hospital, Roermond, Limburg

REFERENCES:
- [Result] Shadid N, Ceulen R, Nelemans P, Dirksen C, Veraart J, Schurink GW, van Neer P, vd Kley J, de Haan E, Sommer A. Randomized clinical trial of ultrasound-guided foam sclerotherapy versus surgery for the incompetent great saphenous vein. Br J Surg. 2012 Aug;99(8):1062-70. doi: 10.1002/bjs.8781. Epub 2012 May 25. PMID 22627969
- [Derived] Lam YL, Lawson JA, Toonder IM, Shadid NH, Sommer A, Veenstra M, van der Kleij AMJ, Ceulen RP, de Haan E, Ibrahim F, van Dooren T, Nieman FH, Wittens CHA. Eight-year follow-up of a randomized clinical trial comparing ultrasound-guided foam sclerotherapy with surgical stripping of the great saphenous vein. Br J Surg. 2018 May;105(6):692-698. doi: 10.1002/bjs.10762. PMID 29652081